CLINICAL TRIAL: NCT03325816
Title: Phase I/II Trial of Anti-PD-1 Checkpoint Inhibitor Nivolumab and 177Lu-DOTA0-Tyr3-Octreotate for Patients With Extensive-Stage Small Cell Lung Cancer
Brief Title: Nivolumab and 177Lu-DOTA0-Tyr3-Octreotate for Patients With Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Bristol-Myers Squibb (Industry); Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1081
Record Dates: First submitted 2017-10-26; First posted 2017-10-30 (Actual); Results first posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Small Cell Lung Cancer; Small Cell Lung Cancer Extensive Stage
Keywords: nivolumab; 177Lu-DOTA0-Tyr3-Octreotate; Lutathera
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Nivolumab; lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase II - Arm 1 (Experimental): Nivolumab will be administered 240mg every 2 weeks. Nivolumab will be given until progressive disease, patient withdrawal, or toxicities.
  The Phase II dose of 177Lu-DOTA0-Tyr3-Octreotate will be the maximum tolerated dose as determined in the Phase I portion.
  Interventions: Drug: Nivolumab; Radiation: 177Lu-DOTA0-Tyr3-Octreotate
- Phase I - Dose Level -1 (Experimental): Nivolumab will be administered 240mg every 2 weeks. Nivolumab will be given until progressive disease, patient withdrawal, or toxicities.
  177Lu-DOTA0-Tyr3-Octreotate dose will be 3.7 GBq (100 mCi) every 8 weeks for 4 doses.
  Interventions: Drug: Nivolumab; Radiation: 177Lu-DOTA0-Tyr3-Octreotate
- Phase I - Dose Level 0 (Experimental): Nivolumab will be administered 240mg every 2 weeks. Nivolumab will be given until progressive disease, patient withdrawal, or toxicities.
  177Lu-DOTA0-Tyr3-Octreotate dose will be 7.4 GBq (200 mCi) every 8 weeks for 4 doses.
  Interventions: Drug: Nivolumab; Radiation: 177Lu-DOTA0-Tyr3-Octreotate
- Phase II - Arm 2 (No Intervention): Patients randomized to this arm will be followed (observation). Cross-over to Phase II Arm 1 at the time of disease progression will be allowed

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is administered intravenously
  Other Names: BMS-936558; Opdivo
  Arms: Phase I - Dose Level -1; Phase I - Dose Level 0; Phase II - Arm 1
Radiation: 177Lu-DOTA0-Tyr3-Octreotate — 177Lu-DOTA0-Tyr3-Octreotate will be administered every 8 weeks. The first dose of 177Lu-DOTA0-Tyr3-Octreotate will be given two weeks after the first administration of nivolumab. Each dose is infused over 30 minutes. On the day of 177Lu-DOTA0-Tyr3-Octreotate infusion, an intravenous bolus of anti-emetics will be given (suggested options: ondansetron (8 mg), granisetron (3 mg), or tropisetron (5 mg)). Administration of 177Lu-DOTA0-Tyr3-Octreotate may be given one day earlier or delayed up to 1 week due to holidays, inclement weather, conflicts, or similar reasons.
  Concurrent amino acids are given with each dose of 177Lu-DOTA0-Tyr3-Octreotate since co-infusion of amino acids leads to a significant reduction (47%) in the mean radiation dose to the kidneys. The amino acid solution and 177Lu-DOTA0-Tyr3-Octreotate are administered in parallel by peripheral vein infusion
  Other Names: Lutathera
  Arms: Phase I - Dose Level -1; Phase I - Dose Level 0; Phase II - Arm 1

SUMMARY:
This research study is being done to assess the safety and tolerability of study drugs, 177Lu-DOTA0-Tyr3-Octreotate (Lutathera) and nivolumab in subjects with small cell lung cancer or advanced or inoperable neuroendocrine tumor of the lung that has overexpressed somatostatin receptors (SSRT). Lutathera is an investigational radioactive agent that targets tumor cells that express SSRT. Nivolumab is an investigational agent that targets and inhibits a pathway that prevents your immune system from effectively fighting your cancer. The combination of these 2 study drugs is investigational. The term "Investigational" in this context means that the drugs have not been approved for clinical use by the US Food and Drug Administration (FDA).

Giving Lutathera and nivolumab together may increase the effectiveness of this therapy. We first need to find out the highest dose of Lutathera that can be given safely together with nivolumab. This study will be the first study to test giving Lutathera together with nivolumab. Once we have found the highest dose of Lutathera that can be given with nivolumab, we will treat more patients with this combination to determine how effective it is.

The purposes of this study are:

To find the highest doses of Lutathera that can be given with nivolumab without causing severe side effects.

To find out the side effects seen by giving Lutathera at different dose levels with nivolumab.

To determine if the amount of something in your tumor called PD-L1 makes you more likely to have a response to the combination of Lutathera and nivolumab.

DETAILED DESCRIPTION:
The purpose of this project to see if the combination of 177Lu-DOTA0-Tyr3-Octreotate and nivolumab is safe and tolerable, and provides PFS benefit compared to observation alone in the maintenance setting in patients with ES-SCLC and no disease progression after first-line platinum-based chemotherapy.

Treatment will be administered on an outpatient basis. A standard dose-escalation phase I design will be used. Three subjects will be enrolled at each dose level in the absence of DLT.

Selection of the starting dose of 177Lu-DOTA0-Tyr3-Octreotate and nivolumab is based on the results from previous clinical studies with each compound used as single agent and the fact that the combination has not been tested in clinical trials. The first dose of 177Lu-DOTA0-Tyr3-Octreotate will be given two weeks after the first administration of nivolumab. Studies have shown that intravenous administration of amino acids has a renal protective effect [46]. An infusion of amino acids (lysine 2.5% and arginine 2.5% in 1 L 0.9% NaCl; 250 mL/h) will be started 30 minutes before the administration of 177Lu-DOTA0-Tyr3-Octreotate and last 4 hours.

Nivolumab will be administered as a fixed dose of 240 mg as an intravenous infusion over 30 minutes every 2 weeks. Nivolumab will be given until progressive disease, patient withdrawal or toxicities.

The phase II portion will consist of patients with ES-SCLC who completed platinum based standard first-line chemotherapy (e.g. 4-6 cycles of platinum plus etoposide or irinotecan) without disease progression (responders plus stable disease) at the time of initiation of the combination therapy with 177Lu-DOTA0-Tyr3-Octreotate and nivolumab. Eligible patients will then be randomly allocated in two arms: one will be treated with the combination of 177Lu-DOTA0-Tyr3-Octreotate and nivolumab, and the other arm will continue be followed (observation) after completion the standard chemotherapy treatment.

Randomization:

Patients who do not receive radiotherapy after chemotherapy

* The randomization must occur within 6 weeks of the last chemotherapy cycle.
* The study treatment must start within 2 weeks from randomization. Patients who receive radiotherapy (including prophylactic cranial radiation and/or thoracic radiation) after chemotherapy
* The randomization must occur within 9 weeks of the last chemotherapy cycle but at least 2 weeks after completion of radiotherapy.
* The first dose of 177Lu-DOTA0-Tyr3-Octreotate cannot be given within 8 weeks of radiotherapy.

Randomization process:

* Randomization will be stratified according to NETSPOT® PET tumor uptake score (Grade 2, 3 and 4).
* OnCore will be used as statistical center and the randomization algorithm will be developed by the study biostatistician.
* The project management department will be the first point of contact for assessment through email.

Courses are defined as 56 days of dosing. Nivolumab will be given until progressive disease, patient withdrawal, or toxicities. For patients randomized to the observation group, cross-over at the time of disease progression will be allowed, since the primary endpoint is PFS and not OS.

ELIGIBILITY:
Inclusion Criteria:

* Phase I

Patients must have cytologically or histologically confirmed relapsed or refractory extensive-disease small-cell lung cancer (ES-SCLC) or non-progressing ES-SCLC after first line chemotherapy, or advanced or inoperable grade I-II pulmonary NETs.

Patients with tumor tissue uptake during NETSPOT® PET that is equal to or higher than that in normal hepatic tissue (grade ≥2) will be eligible. At the discretion of the principal investigator, patients with SCLC whose tumors have lower levels of uptake than liver during NETSPOT® PET may be eligible for the study.

Patients must have measurable disease by RECIST criteria, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan. See Section 7.1.2 for the evaluation of measurable disease.

Toxicities of prior therapy must be resolved to grade 1 or less as per Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 with the exception of alopecia and grade 2, prior platinum-therapy related neuropathy.

Prior radiotherapy or radiosurgery (including prophylactic cranial radiation and/or thoracic radiation) must have been completed at least 2 weeks prior to randomization.

ECOG performance status of 0-1.

Adequate organ and bone marrow function (hemoglobin > 9 g/dL; absolute neutrophil count > 1.5 x 109/L; platelet counts > 100 x 109/L; serum bilirubin < 2 x ULN; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x ULN or < 5 x ULN if liver metastases; calculated creatinine clearance > 50 mL/min).

Life expectancy of at least 3 months.

Age > 18 years.

Women of childbearing potential (WOCBP) must use avoid pregnancy for 23 weeks after the last dose of investigational drug. Men who are sexually active with WOCBP must avoid pregnancy for 31 weeks after the last dose of investigational drug. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile as well as azoospermic men) are not required to avoid pregnancy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropic [HCG]) within 24 hours prior to the start of the study drug.

Women must not be pregnant or breastfeeding.

Ability to understand and willingness to sign a written informed consent document.

* Phase II

Patients must have cytologically or histologically confirmed ES-SCLC and must not have progressed after first line platinum-based chemotherapy regimen before randomization.

Patients with tumor tissue uptake during NETSPOT® PET that is equal to or higher than that in normal hepatic tissue (grade ≥2) will be eligible. It is recommended that NETSPOT® PET be obtained before initiation of chemotherapy, but NETSPOT® PET obtained during or after completion of chemotherapy could be used for screening purpose.

Patients must have measurable disease by RECIST criteria, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan. See Section 7.1.2 for the evaluation of measurable disease.

Toxicities of prior therapy must be resolved to grade 1 or less as per Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 with the exception of alopecia and grade 2, prior platinum-therapy related neuropathy.

Prior radiotherapy or radiosurgery (including prophylactic cranial radiation and/or thoracic radiation) must have been completed at least 2 weeks prior to randomization.

For patients who do not receive radiotherapy after chemotherapy, the randomization must occur within 6 weeks of the last chemotherapy cycle. The study treatment must start within 2 weeks from randomization. For patients who receive radiotherapy (including prophylactic cranial radiation and/or thoracic radiation) after chemotherapy, the randomization must occur within 9 weeks of the last chemotherapy cycle but at least 2 weeks after completion of radiotherapy and the first dose of 177Lu-DOTA0-Tyr3-Octreotate cannot be given within 8 weeks of radiotherapy.

ECOG performance status of 0-1.

Adequate organ and bone marrow function (hemoglobin > 9 g/dL; absolute neutrophil count > 1.5 x 109/L; platelet counts > 100 x 109/L; serum bilirubin < 2 x ULN; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x ULN or < 5 x ULN if liver metastases; calculated creatinine clearance > 50 mL/min).

Life expectancy of at least 3 months.

Age > 18 years.

Women of childbearing potential (WOCBP) must use avoid pregnancy for 23 weeks after the last dose of investigational drug. Men who are sexually active with WOCBP must avoid pregnancy for 31 weeks after the last dose of investigational drug. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile as well as azoospermic men) are not required to avoid pregnancy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropic [HCG]) within 24 hours prior to the start of the study drug.

Women must not be pregnant or breastfeeding.

Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Phase I

Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.

Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.

Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways.

Patients with human immunodeficiency virus (HIV) infection, or active hepatitis B or C virus infection will be excluded.

Patients who received prior anti-tumoral radionuclide therapy (with unsealed sources) are not eligible for the study.

Prior major surgery within 12 weeks or prior major surgery from which the patient has not sufficiently recovered yet.

Untreated and uncontrolled second tumor in the past 2 years.

Logistical or psychological hindrance to participation in clinical research.

Uncontrolled or significant cardiovascular disease, including any of the following:

* Symptomatic congestive heart failure (New York Heart Association Classification Class II).
* Cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), or unstable angina.
* Uncontrolled hypertension or uncontrolled cardiac arrhythmia.

Any other medical condition that in the Investigator's opinion would not make the patient a good candidate for the study.

* Phase II

Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.

Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.

Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways.

Patients with human immunodeficiency virus (HIV) infection, or active hepatitis B or C virus infection will be excluded.

Patients who received prior anti-tumoral radionuclide therapy (with unsealed sources) are not eligible for the study.

Prior major surgery within 12 weeks or prior major surgery from which the patient has not sufficiently recovered yet.

Untreated and uncontrolled second tumor in the past 2 years.

Logistical or psychological hindrance to participation in clinical research.

Uncontrolled or significant cardiovascular disease, including any of the following:

* Symptomatic congestive heart failure (New York Heart Association Classification Class II).
* Cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), or unstable angina.
* Uncontrolled hypertension or uncontrolled cardiac arrhythmia.

Any other medical condition that in the Investigator's opinion would not make the patient a good candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2020-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chul Kim, MD, Principal Investigator — Georgetown University
Locations (2):
- United States (2):
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim C, Liu SV, Subramaniam DS, Torres T, Loda M, Esposito G, Giaccone G. Phase I study of the 177Lu-DOTA0-Tyr3-Octreotate (lutathera) in combination with nivolumab in patients with neuroendocrine tumors of the lung. J Immunother Cancer. 2020 Jul;8(2):e000980. doi: 10.1136/jitc-2020-000980. PMID 32616557

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I - Dose Level -1: Nivolumab will be administered 240mg every 2 weeks, intravenously until progressive disease, patient withdrawal, or toxicities. 177Lu-DOTA0-Tyr3-Octreotate dose will be 3.7 GBq (100 mCi), infused over 30 minutes, every 8 weeks for 4 doses. The first dose of 177Lu-DOTA0-Tyr3-Octreotate will be given two weeks after the first administration of nivolumab and an intravenous bolus of anti-emetics will be given. Concurrent amino acids are given in parallel by peripheral vein infusion with each dose of 177Lu-DOTA0-Tyr3-Octreotate.
- Phase I - Dose Level 0: Nivolumab will be administered 240mg every 2 weeks, intravenously until progressive disease, patient withdrawal, or toxicities. 177Lu-DOTA0-Tyr3-Octreotate dose will be 7.4 GBq (200 mCi), infused over 30 minutes, every 8 weeks for 4 doses. The first dose of 177Lu-DOTA0-Tyr3-Octreotate will be given two weeks after the first administration of nivolumab and an intravenous bolus of anti-emetics will be given. Concurrent amino acids are given in parallel by peripheral vein infusion with each dose of 177Lu-DOTA0-Tyr3-Octreotate.
Period: Overall Study
Arm/Group | Phase I - Dose Level -1 | Phase I - Dose Level 0
Started | 3 | 6
Completed | 3 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I - Dose Level -1 | Phase I - Dose Level 0 | Total
Number analyzed (Participants) | 3 | 6 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 5 | 6
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 5
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 6 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 1 | 6 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase I - Recommended Phase II Dose (RP2D) of 177Lu-DOTA0-Tyr3-Octreotate
Description: Maximum tolerated dose of 177Lu-DOTA0-Tyr3-Octreotate as determined during the phase I portion.
Time Frame: 12 months
Measure: Number; unit: GBq
Groups:
- Phase I: Nivolumab will be administered 240mg every 2 weeks, intravenously until progressive disease, patient withdrawal, or toxicities. 177Lu-DOTA0-Tyr3-Octreotate dose will be 3.7 or 7.4 GBq (200 mCi), infused over 30 minutes, every 8 weeks for 4 doses. The first dose of 177Lu-DOTA0-Tyr3-Octreotate will be given two weeks after the first administration of nivolumab and an intravenous bolus of anti-emetics will be given. Concurrent amino acids are given in parallel by peripheral vein infusion with each dose of 177Lu-DOTA0-Tyr3-Octreotate.
Arm/Group | Phase I
Number analyzed (Participants) | 9
GBq | 7.4

2. Primary Outcome: Phase II - Progression Free Survival
Description: Time between start of treatment and tumor progression or death
Time Frame: 12 months
Population: Phase II outcome- analysis not applicable. Phase II not started per Sponsor decision.
Groups:
- Phase II: Nivolumab will be administered 240mg every 2 weeks, intravenously until progressive disease, patient withdrawal, or toxicities. 177Lu-DOTA0-Tyr3-Octreotate dose will be 7.4 GBq (200 mCi), infused over 30 minutes, every 8 weeks for 4 doses. The first dose of 177Lu-DOTA0-Tyr3-Octreotate will be given two weeks after the first administration of nivolumab and an intravenous bolus of anti-emetics will be given. Concurrent amino acids are given in parallel by peripheral vein infusion with each dose of 177Lu-DOTA0-Tyr3-Octreotate.
Arm/Group | Phase II
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Treatment Related Adverse Events
Description: Adverse events and serious adverse events experienced by subjects
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Dose Level -1 | Phase I - Dose Level 0
Number analyzed (Participants) | 3 | 6
Participants | 3 | 6

4. Secondary Outcome: Phase II - Overall Survival
Description: Time between start of treatment and death
Time Frame: 24 months
Population: Phase II outcome- analysis not applicable. Phase II not started per Sponsor decision.
Arm/Group | Phase II
Number analyzed (Participants) | 0

5. Secondary Outcome: Phase II - Disease Control Rate
Description: The percentage of patients who achieve complete response, partial response and stable disease
Time Frame: 12 months
Population: Phase II outcome- analysis not applicable. Phase II not started per Sponsor decision.
Arm/Group | Phase II
Number analyzed (Participants) | 0

6. Secondary Outcome: Phase II - Objective Response Rate
Description: The proportion of patients with tumor size reduction
Time Frame: 12 months
Population: Phase II outcome- analysis not applicable. Phase II not started per Sponsor decision.
Arm/Group | Phase II
Number analyzed (Participants) | 0

7. Secondary Outcome: Phase II - Metabolic Response
Description: As measured by NETSPOT PET scan
Time Frame: 12 months
Population: Phase II outcome- analysis not applicable. Phase II not started per Sponsor decision.
Arm/Group | Phase II
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Phase I - Dose Level -1 | Phase I - Dose Level 0
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Dose Level -1 (N=3) | Phase I - Dose Level 0 (N=6)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Biliary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) — Ascending Cholangitis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Dose Level -1 (N=3) | Phase I - Dose Level 0 (N=6)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (2)
Bladder Spasm (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchial Infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Edema Limbs (General disorders) | 1 (1) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (3) | 2 (4)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (4)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (4)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 4 (6)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Eczema (Psoriasis)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3)
Weight Loss (Investigations) | 1 (1) | 1 (1)
General disorders and administration site conditions Other, specify (General disorders) | 0 (0) | 1 (1) — Night sweats
General disorders and administration site conditions Other, specify (General disorders) | 0 (0) | 1 (1) — Slurred speech
General disorders and administration site conditions Other, specify (General disorders) | 0 (0) | 1 (1) — Transaminitis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT03325816/Prot_SAP_001.pdf